CLINICAL TRIAL: NCT04705519
Title: A Prospective, Non-randomized, Multicenter, Phase II Study of Nab-paclitaxel Combined with Bevacizumab for Unresectable Recurrent or Metastatic Extrapulmonary Neuroendocrine Carcinoma
Brief Title: Nab-paclitaxel Combined with Bevacizumab in the Treatment of Metastatic Extrapulmonary Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGOG3006/NEC-BEVAX
Record Dates: First submitted 2021-01-06; First posted 2021-01-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-09

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nab-paclitaxel Combined With Bevacizumab (Experimental): Nab-paclitaxel, Bevacizumab
  Interventions: Drug: Nab-paclitaxel Combined With Bevacizumab

INTERVENTIONS:
Drug: Nab-paclitaxel Combined With Bevacizumab — Nab-paclitaxel 150mg/m2 ，iv drip, d1, Bevacizumab 5mg/kg, iv drip, d1, q2w.

SUMMARY:
This is an open-label, phase II study evaluating efficacy and safety of Nab-paclitaxel Combined With Bevacizumab for unresectable Recurrent or metastatic extrapulmonary neuroendocrine carcinoma.

DETAILED DESCRIPTION:
Nab-paclitaxel Combined With Bevacizumab will be evaluated in participants who have had ≥ 1 line of previous treatment. The primary endpoint is the Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provided written informed consent to be subjects in this trial
2. Aged ≥18 years
3. Has histologically-confirmed diagnosis of locally advanced unresectable or metastatic extrapulmonary neuroendocrine carcinoma
4. Has received and progressed on ≥1 prior systemic therapy for their advanced disease.
5. Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
6. Have measurable disease as defined by RECIST 1.1 as determined by investigator assessment
7. Agree to provide tumor tissue sample deemed adequate for histopathology confirmation
8. Adequate Organ Function Laboratory Values:

   Hemoglobin ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelets ≥80×109/L; AST and ALT ≤ 1.5 ULN or ≤ 3 ULN for subjects with liver metastases; Total bilirubin ≤1.5 ULN; Serum creatinine ≤1.5 ULN or measured or calculated creatinine clearance > 50ml/min; Albumin ≥ 30g/L;
9. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication and must be willing to use an adequate method of contraception for the course of the study through 90 days after the last dose of study medication. Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy

Exclusion Criteria:

1. Patients have recovered adverse events associated with pretreatment to Grade 1 or lower with CTCAE v5.0 excluding alopecia
2. Patients have an active malignancy (except for definitively treated basal cell carcinoma of the skin, or carcinoma-in-situ of the cervix) within the past 5 years
3. Patients with uncontrolled central nervous system metastasis
4. Received anti-tumor therapy within 4 weeks, including: chemotherapy (the washout period of oral fluorouracil drugs is 2 weeks), targeted therapy (the washout period of small molecule targeted drugs is 2 weeks or 5 half-lives, whichever is shorter), immunotherapy, etc.;
5. Received radical radiotherapy (including >25% bone marrow radiotherapy) and brain radiotherapy within 4 weeks; brachytherapy (such as implantation of radioactive particles) within 60 days; received palliative radiotherapy for bone metastases within 1 week;
6. Patients with a history of prior treatment with docetaxel, paclitaxel, nab-paclitaxel or bevacizumab
7. Received surgery within 4 weeks or unhealed wounds, Ulcers, fractures;
8. Uncontrollable malignant pleural effusion, ascites, or pericardial effusion (defined as the investigator's judgment cannot be effectively controlled by diuretics or puncture);
9. Patients have gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresected tumors, or other conditions judged that may cause gastrointestinal bleeding or perforation;
10. Patients with evidence or medical history of thrombosis or obvious bleeding tendency within 2 months (bleeding> 30 mL within 2 months, hematemesis, melena, blood in the stool), hemoptysis (> 5 mL of fresh blood within 4 weeks);
11. Patients have arterial thrombosis or deep vein thrombosis occurred within 6 months; or stroke and/or transient ischemic attack occurred within 12 months;
12. Active heart disease that is not well controlled, e.g. symptomatic coronary heart disease, New York Heart Association (NYHA) congestive heart failure of grade II or above, severe arrhythmias requiring drug intervention, myocardial infarction within the past 6 months, LVEF<50%
13. Patients judged with clinically significant electrolyte abnormalities
14. Patients have an active infection or an unexplained fever (temperature> 38.5℃) during the screening period or before the first administration
15. Patients with active tuberculosis (TB) who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year
16. Is pregnant or breastfeeding
17. Patients were judged unsuitable as subjects of this trial by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | an expected average of 24 months
  Duration from the date of initial treatment to the date of death due to any cause

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
Duration of Response (DoR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The percentage of patients who achieve complete remission(CR) or partial remission (PR) or stable disease(SD) determined by the RECIST v1.1 criteria.
Progression Free Survival (PFS) | an expected average of 24 months
  A duration from the date of initial treatment to radiographic disease progression or death of any cause
Disease Control Rate (DCR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Proportion of objective complete response, partial response and stable patients
Adverse events | an expected average of 24 months
  Including other occasional or rare AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang P, Li S, Jia R, Hao J, Chen C, Gan S, Li J, Shen L, Lu M. Nab-paclitaxel plus bevacizumab for patients with metastatic extrapulmonary neuroendocrine carcinoma: a phase 2 single-arm study. EClinicalMedicine. 2025 Oct 24;90:103598. doi: 10.1016/j.eclinm.2025.103598. eCollection 2025 Dec. PMID 41209655